CLINICAL TRIAL: NCT07330167
Title: Does Boredom With Simultaneously Perceived Pain Affect Sensitivity to Pressure and Other Pain-related Variables?
Brief Title: Does Boredom With Simultaneously Perceived Pain Affect Pressure Pain Thresholds
Acronym: BPPPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Helena Gunnarsson, Dr, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr 2025-06262-01; Linnaeus University (Other: Linnaeus University)
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pain Thresholds
Keywords: Pressure Pain Thresholds; Pain; Emotions
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Within-subjects design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Boredom intervention (Experimental): The participant will watch a short video ( boredom) 2.30 minutes in length while experimental pain is induced.
  Interventions: Other: Boredom intervention
- Humorous control intervention (Active Comparator): The participant will watch a short humorous video 2.30 minutes in length while experimental pain is induced.
  Interventions: Other: Humorous
- Control intervention (No Intervention): The participant will wait for 2.30 minutes with experimentally induced pain.

INTERVENTIONS:
Other: Boredom intervention — A short boring video will be shown.
  Other Names: Emotional
  Arms: Boredom intervention
Other: Humorous — A short humorous video will be shown.
  Arms: Humorous control intervention

SUMMARY:
The purpose of this study is to investigate if different emotional states such as boredom and happiness could influence mechanical pain thresholds and other pain - related variables such as pain tolerance, pain intensity and pain - related negative affect.

DETAILED DESCRIPTION:
Participants will be randomized into 3 different groups watching different short video-clips (2.30 min), while at the same time experience short-lasting, experimentally induced pain. The boredom emotions group will watch a short boring video, the positive emotions group will watch a video containing a stand-up comedy show and this video will also be the distraction control, and the control group will just wait for 2.30 min, without any instructions about what to think about. Pressure pain thresholds will be measured with an algometer before and after the video-clip combined with experimental pain interventions.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age and below 80 years of age.
* Fluent in Swedish.

Exclusion Criteria:

* Pain anywhere in the body during the test session.
* Known neurological disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold | The Pressure Pain Thresholds will be measured directly after the intervention.
  Pressure Pain Thresholds will be measured with a handheld algometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Helena Gunnarsson, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided